CLINICAL TRIAL: NCT03354676
Title: Adiponectin, Leptin, h-CRP Values in Obese Children - Important Markers for Metabolic Syndrome?
Acronym: ChildObes
Status: Completed | Type: Observational
Sponsor: Alexandru Florin Rogobete (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Sponsor-Investigator, Alexandru Florin Rogobete, MSc, PhDs, Clinical Researcher, Romanian Society of Anesthesia and Intensive Care
Organization: Romanian Society of Anesthesia and Intensive Care (Other)
Other Study IDs: 12870
Record Dates: First submitted 2017-09-12; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Obesity, Metabolically Benign
Keywords: adipokines, metabolic syndrome, obese children
MeSH Terms: conditions — Obesity, Metabolically Benign; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MetS+: Obese group with metabolic syndrome/Data processing from Patient Medical Files
  Interventions: Other: MetS+
- MetS-: Obese group without metabolic syndrome/Data processing from Patient Medical Files
  Interventions: Other: MetS-

INTERVENTIONS:
Other: MetS+ — Data processing from Patient Medical Files
  Groups: MetS+
Other: MetS- — Data processing from Patient Medical Files
  Groups: MetS-

SUMMARY:
Obesity is a chronic inflammatory disorder in which leptin, adiponectin and C reactive protein (CRP) play an important role. This study aimed to investigate the relationship between markers of adiposity like leptin, adiponectin and high sensitive C reactive protein (hsCRP) in obese children, and to determine whether these adipokines are significant markers in defining metabolic syndrome in pediatric population

DETAILED DESCRIPTION:
The idea that adipose tissue is just a form of energy storage has changed dramatically in recent years. Currently, adipose tissue is considered to be a true endocrine gland that fulfills multiple roles in regulating different biological functions. Communication between adipose tissue and the rest of the systems is accomplished through bioactive mediators (adipokines) Adipokines control energy homeostasis and are involved in metabolic, endocrine and immunological processes.This study aimed to investigate the relationship between markers of adiposity like leptin, adiponectin and high sensitive C reactive protein (hsCRP) in obese children, and to determine whether these adipokines are significant markers in defining metabolic syndrome in pediatric population.The current retrospective observational study was conducted at the "Louis Turcanu" Emergency Hospital Timisoara over a period of one year, from July 2013 and June 2014. All inborn patient files were analyzed as anonymised limited data sets from archived records of the Endocrinology, Diabetology and Cardiology department.

ELIGIBILITY:
Inclusion Criteria:

* obese children (BMI> 95th percentile)

Exclusion Criteria:

* obesity caused by endocrine disease, syndromic obesity, systemic disease or acute illness.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children admitted to the Endocrinology, Diabetology and Cardiology Department who met the Inclusion Criteria
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Defining obesity in the pediatric population | Weight and height were measured on day 1 of admission. Obesity was defined as a BMI > the 95th percentile.
  Measuring weight in kilograms and height in meters in order to calculate BMI and represent it on the percentile graph.
Leptin changes in the obese children with metabolic syndrome | Leptin levels were measured on day 1 of admission. Normal range was considered < 24ng/ml.
  Evaluating leptin in the obese group with metabolic syndrome
Adiponectin changes in the obese children with metabolic syndrome | Adiponectin levels were measured on day 1 of admittance in children aged between 4 and18 years. Levels 4-26 mcg/ml were defined as normal values.
  Evaluating adiponectin in the obese group with metabolic syndrome
Assessing cardiovascular risk in the obese children with metabolic syndrome | hsCRP levels were measured on day 1 of admittance in children aged between 4 and 18 years. Normal levels were considered between 0.1-2.8 mg/l
  Evaluating hsCRP in the obese group with metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Florin Rogobete, PhDS, Principal Investigator — Romanian Society of Anesthesia and Intensive Care

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyazit F, Unsal MA. Obesity and insulin resistance are significant predictors of serum leptin levels. J Turk Ger Gynecol Assoc. 2017 Sep 1;18(3):158-159. doi: 10.4274/jtgga.2017.0027. No abstract available. PMID 28890432
- [Background] Lopez-Quintero A, Garcia-Zapien AG, Flores-Martinez SE, Diaz-Burke Y, Gonzalez-Sandoval CE, Lopez-Roa RI, Medina-Diaz E, Munoz-Almaguer ML, Sanchez-Corona J. Contribution of polymorphisms in the LEP, LEPR and RETN genes on serum leptin and resistin levels in young adults from Mexico. Cell Mol Biol (Noisy-le-grand). 2017 Aug 30;63(8):10-18. doi: 10.14715/cmb/2017.63.8.3. PMID 28886308
- [Background] Bagherniya M, Khayyatzadeh SS, Heidari Bakavoli AR, Ferns GA, Ebrahimi M, Safarian M, Nematy M, Ghayour-Mobarhan M. Serum high-sensitive C-reactive protein is associated with dietary intakes in diabetic patients with and without hypertension: a cross-sectional study. Ann Clin Biochem. 2018 Jul;55(4):422-429. doi: 10.1177/0004563217733286. Epub 2017 Nov 23. PMID 28882065